CLINICAL TRIAL: NCT02772185
Title: Neurostimulation and Cognitive Intervention in Alzheimer's Disease
Acronym: NeuroAD
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Suellen Marinho Andrade, Professor, Federal University of Paraíba
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NeuroAD
Record Dates: First submitted 2016-05-05; First posted 2016-05-13 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- active tDCS plus real CT (Experimental): Participants will receive active transcranial direct current stimulation and real cognitive training.
  Interventions: Device: active tDCS; Behavioral: real CT
- sham tDCS plus real CT (Experimental): Participants will receive sham transcranial direct current stimulation and real cognitive training.
  Interventions: Device: sham tDCS; Behavioral: real CT
- active tDCS plus placebo CT (Experimental): Participants will receive active transcranial direct current stimulation and placebo cognitive training.
  Interventions: Device: active tDCS; Behavioral: placebo CT
- sham tDCS plus placebo CT (Placebo Comparator): Participants will receive sham transcranial direct current stimulation and placebo cognitive training.
  Interventions: Device: sham tDCS; Behavioral: placebo CT

INTERVENTIONS:
Device: active tDCS — Duration: 30 minutes; Intensity: 2 mA; Placement:left and right parietal cortex, left and right DLPFC, left inferior frontal gyrus and left superior temporal gyrus
  Arms: active tDCS plus placebo CT; active tDCS plus real CT
Device: sham tDCS — The procedure is the same as for active tDCS, but the in the placebo tDCS the stimulation is non-active / sham.
  Arms: sham tDCS plus placebo CT; sham tDCS plus real CT
Behavioral: real CT — Cognitive tasks designed to relate to the region of the brain being stimulated (left and right parietal cortex, left and right DLPFC, left inferior frontal gyrus and left superior temporal gyrus).
  Arms: active tDCS plus real CT; sham tDCS plus real CT
Behavioral: placebo CT — Videos (short films) will be presented during the neurostimulation
  Arms: active tDCS plus placebo CT; sham tDCS plus placebo CT

SUMMARY:
This study is a double blind, sham-controlled clinical trial aiming to compare the long-term effects of stimulation in Alzheimer's Disease (AD). Sixty early AD patients will take part in a phase II/III clinical study over a 1-year period. The study involves transcranial direct current stimulation (tDCS), cognitive training (CT), detailed neuropsychological and neurological testing. These assessments will occur at baseline, then again at two month (end point). Those who achieve clinical improvement with neurostimulation and cognitive therapy will be invited to receive treatment for 12 months as part of a follow-up study.

DETAILED DESCRIPTION:
The patients will be randomized into 1 of 4 groups: active tDCS plus real CT, active tDCS plus placebo CT, sham tDCS plus real CT, sham tDCS plus placebo CT. Each group will receive treatment for 30 minutes a day, 3 days a week for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 60-90 years
* Patients diagnosed with Alzheimer's Disease, according to the DSM-IV (Diagnostic and Statistical Manual of Mental Disorders) and NINCDS-ADRDA (National Institute for Communicative Disorders and Stroke - Alzheimer's Disease and Related Disorders Association) criteria
* Score between 18 and 26 on the Mini Mental State Examination
* Have a CDR (Clinical Dementia Rating) of 1.0
* If medicated for AD, then use of cholinesterase inhibitors, for at least 3 months and on stable dose for at least 60 days prior to screening.

Exclusion Criteria:

* Pre-existing structural brain abnormalities,
* Other neurologic or psychiatric diagnoses
* Transcranial direct current stimulation criteria: patients with implanted metallic or electronic devices; pacemaker; seizures; pregnancy; any other condition that might limit or interfere in the sensorimotor system

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-05; Primary Completion 2018-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Change in cognitive function assessed on the Alzheimer's Disease Assessment Scale-cognitive subscale (ADAS-Cog) | Baseline (week 1), Endpoint (week 8) and Follow up (assessed up to 12 months)

SECONDARY OUTCOMES:
Change in cognitive ability assessed on the Wechsler Adult Intelligence Scale | Baseline (week 1), Endpoint (week 8) and Follow up (assessed up to 12 months)
Change in visuo-spatial working memory assessed on the Corsi block task | Baseline (week 1), Endpoint (week 8) and Follow up (assessed up to 12 months)
Change in verbal working memory assessed on the Digit Span task | Baseline (week 1), Endpoint (week 8) and Follow up (assessed up to 12 months)
Change in speed of cognitive processing and executive functioning assessed on the Trail Making Test | Baseline (week 1), Endpoint (week 8) and Follow up (assessed up to 12 months)
Change in executive function assessed on the Stroop Color and Word Test | Baseline (week 1), Endpoint (week 8) and Follow up (assessed up to 12 months)
Change in verbal fluency assessed on the FAS Verbal Fluency Test | Baseline (week 1), Endpoint (week 8) and Follow up (assessed up to 12 months)
Change in functional ability assessed on the Disability Assessment Dementia | Baseline (week 1), Endpoint (week 8) and Follow up (assessed up to 12 months)
Change in visual recognition assessed on the Poppelreuter-Ghent's Overlapping Figures test | Baseline (week 1), Endpoint (week 8) and Follow up (assessed up to 12 months)
Change in behavioral and psychological disturbances assessed on the Neuropsychiatric Inventory Questionnaire | Baseline (week 1), Endpoint (week 8) and Follow up (assessed up to 12 months)
Change in subjective burden among caregivers assessed on the Zarit Burden Interview | Baseline (week 1), Endpoint (week 8) and Follow up (assessed up to 12 months)
Change in electrical activity of the brain assessed on the Electroencephalogram (EEG) | Baseline (week 1), Endpoint (week 8) and Follow up (assessed up to 12 months)
Side Effects Questionnaire | From date of first neurostimulation until the date of last neurostimulation, assessed up to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Suellen Andrade, João Pessoa, Paraíba, Brazil

REFERENCES:
- [Derived] Andrade SM, da Silva-Sauer L, de Carvalho CD, de Araujo ELM, Lima EO, Fernandes FML, Moreira KLAF, Camilo ME, Andrade LMMDS, Borges DT, da Silva Filho EM, Lindquist AR, Pegado R, Morya E, Yamauti SY, Alves NT, Fernandez-Calvo B, de Souza Neto JMR. Identifying biomarkers for tDCS treatment response in Alzheimer's disease patients: a machine learning approach using resting-state EEG classification. Front Hum Neurosci. 2023 Oct 4;17:1234168. doi: 10.3389/fnhum.2023.1234168. eCollection 2023. PMID 37859768
- [Derived] Marchi LZ, Ferreira RGD, de Lima GNS, da Silva JAS, da Cruz DMC, Fernandez-Calvo B, Andrade SMMDS. Multisite transcranial direct current stimulation associated with cognitive training in episodic memory and executive functions in individuals with Alzheimer's disease: a case report. J Med Case Rep. 2021 Apr 22;15(1):185. doi: 10.1186/s13256-021-02800-x. PMID 33883015
- [Derived] Andrade SM, de Oliveira EA, Alves NT, Dos Santos ACG, de Mendonca CTPL, Sampaio DDA, da Silva EEQC, da Fonseca EKG, de Almeida Rodrigues ET, de Lima GNS, Carvalho J, da Silva JAS, Toledo M, da Rosa MRD, Gomes MQC, de Oliveira MM, Lemos MTM, Lima NG, Inacio P, da Cruz Ribeiro E Rodrigues PM, Ferreira RGD, Cavalcante R, de Brito Aranha REL, Neves R, da Costa E Souza RM, Portugal TM, Martins WKN, Pontes V, de Paiva Fernandes TM, Contador I, Fernandez-Calvo B. Neurostimulation Combined With Cognitive Intervention in Alzheimer's Disease (NeuroAD): Study Protocol of Double-Blind, Randomized, Factorial Clinical Trial. Front Aging Neurosci. 2018 Nov 2;10:334. doi: 10.3389/fnagi.2018.00334. eCollection 2018. PMID 30450044